CLINICAL TRIAL: NCT03750474
Title: Comparison of the Stiffness of the Lumbar Back Muscles Between Low Back Pain and Healthy Controls Using Magnetic Resonance Elastography and Shear Wave Elastography
Brief Title: Comparison of the Stiffness of the Lumbar Back Muscles Between Low Back Pain and Healthy Controls
Acronym: PARA-ELASTO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: K180403J; 2017-A02799-44 (Other: IDRCB)
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Low Back Pain
Keywords: elastography; magnetic resonance imaging
MeSH Terms: conditions — Low Back Pain | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient with chronic low back pain (Experimental): magnetic resonance elastography and shear wave elastography of the back muscles
  Interventions: Diagnostic Test: magnetic resonance elastography and shear wave elastography
- healthy controls (Other): magnetic resonance elastography and shear wave elastography of the back muscles
  Interventions: Diagnostic Test: magnetic resonance elastography and shear wave elastography

INTERVENTIONS:
Diagnostic Test: magnetic resonance elastography and shear wave elastography — magnetic resonance elastography and shear wave elastography of the back muscles

SUMMARY:
Chronic low back pain remains a major public health issue. Low back pain is frequently associated with stiffness changes of the lumbar back muscles. The techniques which assess the stiffness of the back muscles are poorly reliable and do not allow the quantification of stiffness changes. Elastography (magnetic resonance imaging and ultrasound) can be used to objectively and non-invasively quantify in vivo tissue elasticity. The aim of the investigator's study is to compare the stiffness in the main lumbar back muscles (i.e. the erector spinae and the multifidus) by using magnetic resonance elastography and shear wave elastography.

DETAILED DESCRIPTION:
"Chronic low back pain (CLBP) is commonly associated with increased trunk stiffness detected by quick release methods and motion track systems as well as increased back muscles stiffness identified by manual palpatory procedures or strain elastography. However, these techniques are qualitative and operator dependent, hence they remain poorly reliable.

Over the last decade, imaging techniques have become very helpful to characterize the biomechanical properties of tissues in vivo. Today, supersonic shear wave elastography (SWE) allows real time mapping of the elastic shear modulus. Also, magnetic resonance allows mapping and quantifying stiffness within a large volume of tissue. Elastography is efficient in the characterization of passive and active muscle forces, in highlighting the influence of muscle stiffness on joint stiffness and in showing stiffness changes related to muscle diseases Imaging plays a key role in the management of CLBP; It allows to reach specific radiological diagnosis such as tumor, inflammatory, or arthritis. However, in many cases, MRI did not find a specific cause to low back pain and the low back pain is reported as "non-specific". Myofascial disorders are also responsible for non-specific CLBP.

The main objective of this study is to compare the shear modulus of the main lumbar back muscles (erector spinae and multifidus) between patients with low back pain and healthy controls.

Second objectives are to assess: the relationship between the stiffness of the back muscles and clinical stiffness, the influence of age and sex on the elasticity of the back muscles, the relationship between the surface of the paravertebral muscles and the elasticity; the relationship between the elasticity of the hypaxial muscles (in front of the spine) and the epaxial muscles (behind the spine =back muscles), the relationship between fatty infiltration and elasticity of the back muscles, the relationship between inflammation / edema of back muscles and stiffness of the back muscles, the influence of the muscular stretching on the elasticity of the paravertebral muscles, the difference of elasticity in the direction of the muscle fibers (oblique coronal) and perpendicular (axial), the stiffness difference the between the right and left muscles, the role of different postures on muscle elasticity, the relationship between the elasticity of the back muscles and the intensity and type of pain, the relationship between the elasticity of the paravertebral muscles and disco-vertebral and / or posterior apophyseal pathology.

The inclusion of 26 patients and 26 controls will demonstrate a difference in mean elasticity modulus of 1.1 standard deviation (between patients and controls), with 90% and an alpha risk of 5%.

Patients will undergo an MRI (sagittal Short Inversion Time Inversion Recovery (STIR) and T1, coronal STIR and axial T1) in the management of low back pain. At the end of their examination, two elastography-sequences will be performed (axial and coronal plane). After the MRI, the patient will undergo a shear wave sonoelastography.

Healthy controls will undergo an MRI (sagittal T1 and T2) and two elastography-sequences (axial and coronal plane). After the MRI, the patient will undergo a an shear wave sonoelastography .

Healthy controls will be recruited in the hospital and university. Patients will be included when the appointment for MRI was made. Signed informant consent will be obtained after oral and written information.

The data manager will be trained to complete the case report form (CRF) and questionnaires; CRF and questionnaire. The entries that are not done according to procedure will result in inaccurate research data and inadequate source documentation. All data collected in the CRF will be scanned in a timely manner, then saved in an Exel folder, and initialized and dated by the data manager. Scanned data will be saved to the local database and on Universal Serial Bus (USB) disk. Computers designated for data entry, export and scanning will be password protected.

Data reported as missing, unavailable, non-reported, uninterpretable, or considered missing because of data inconsistency or out-of-range results were excluded.

Descriptive and comparative statistics will be done. The shear modulus will be compared between cases and controls using a Student's test (or Wilcoxon's test). For the secondary criteria, the comparison between qualitative variables will be made using the Chi² test, the comparison between a quantitative variable and a qualitative variable with a Student test (or Wilcoxon) or a one-way analysis of variance ( or Kruskal-Wallis test), the association between quantitative variables with the calculation of the Pearson (or Spearman) coefficient, depending on the conditions of application.

ELIGIBILITY:
Inclusion criteria for patient

* Chronic low back pain (defined as low back pain for more than 3 months)
* Lumbar MRI without planned injection in chronic low back pain assessment
* Age between 18 and 80 years
* Ability to keep still in an MRI machine
* No contraindication to MRI
* No major sporting activity within 48 hours prior to the exam
* Informed and written consent"

Inclusion criteria for Health control

* No lumbar pain symptomatology, no lumbar static disorder, known neuromuscular pathology
* Age between 18 and 80 years
* Ability to keep still in an MRI machine
* No contraindication to MRI
* Informed and written consent

Exclusion criteria

* Inability to keep still in an MRI machine
* Intercurrent illness that may interfere with exam results
* Concomitant use of medications that may alter muscle metabolism
* Need to inject contrast during MRI
* Non-affiliation to a social security
* Minors, protected adults, persons unable to consent, persons under the protection of justice

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Stiffness mapping and measurement of the shear modulus (m/s) in the multifidus and the erector spinae (1) with magnetic resonance elastography (Aera; 1,5T) | 18 months
  First, the subjects undergoes a magnetic resonance elastography in decubitus in two postures: at rest and with stretching of back muscles (hip flexion). Then, stiffness will be measurement with sonography in several postures: prone position, upright, bending forward, bending backward.

CONTACTS AND LOCATIONS:
Overall Officials: Maud CREZE, PHU, Principal Investigator — APHP
Locations (1):
- Hopital Bicêtre - Radiology Department, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No